CLINICAL TRIAL: NCT00869323
Title: Phase II Trial of Bortezomib and Rituximab for Patients With Post Transplant Lymphoproliferative Disorders (PTLD)
Brief Title: Bortezomib and Rituximab in Treating Patients With Post-Transplant Lymphoproliferative Disorders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008LS043; MT2008-05R (Other: Blood and Marrow Transplantation Program); 0806M37121 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Lymphoproliferative Disorder
Keywords: post-transplant lymphoproliferative disorder
MeSH Terms: conditions — Lymphoproliferative Disorders | interventions — Rituximab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated Patients (Experimental): This group includes patients receiving Bortezomib and Rituximab for post-transplant lymphoproliferative disorders (PTLD).
  Interventions: Biological: rituximab; Drug: bortezomib

INTERVENTIONS:
Biological: rituximab — 375 mg/m^2 intravenously on Days 1,8, 15 and 22
  Other Names: Rituxan
Drug: bortezomib — 1.3 mg/m^2 intravenous bolus days 1, 8, 15 and 22
  Other Names: Velcade

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Monoclonal antibodies, such as rituximab, can block cancer cell growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving bortezomib together with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with rituximab works in treating patients with post-transplant lymphoproliferative disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the overall (complete and partial) response rates in patients with CD20+ post-transplant lymphoproliferative disorders treated with bortezomib and rituximab.

Secondary

* To evaluate the duration of remission, time to treatment failure, relapse-free survival, and overall survival of these patients.
* To characterize the quantitative and qualitative toxicities of this regimen.

OUTLINE:

* Induction therapy: Patients receive bortezomib intravenously (IV) and rituximab IV on days 1, 8, 15, and 22.

Patients achieving complete remission (CR) after completion of induction therapy proceed to maintenance therapy after 6 months of rest. Patients achieving partial remission (PR) or stable disease after completion of induction therapy receive additional bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR/PR after completion of bortezomib therapy proceed to maintenance therapy after 3 months of rest.

* Maintenance therapy: Patients receive bortezomib IV and rituximab IV on days 1, 8, 15, and 22. Treatment repeats every 6 months for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20+ B-cell post-transplant lymphoproliferative disorder
* Has undergone prior solid organ transplant
* Measurable disease as defined by Non-Hodgkin Lymphoma Response Criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1,000/mm³
* Platelet count ≥ 75,000/mm³
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 40 mL/min
* Alanine transaminase (ALT) and Aspartate aminotransferase (AST) ≤ 3 times upper limit of normal
* Total bilirubin ≤ 2.0 mg/dL

Exclusion Criteria:

* Pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Peripheral neuropathy ≥ grade 2
* Known lymphomatous meningitis or central nervous system (CNS) involvement
* HIV infection
* Uncontrolled infection
* Myocardial infarction within the past 6 months or uncontrolled angina
* New York Heart Association class III-IV heart failure
* Severe uncontrolled ventricular arrhythmias
* Evidence of acute ischemia or active conduction system abnormalities by electrocardiogram (EKG)
* Concurrent serious medical or psychiatric disorder (e.g., active infection or uncontrolled diabetes) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study
* Diagnosis or treatment for another malignancy within the past 3 years, except completely resected basal cell carcinoma or squamous cell carcinoma of the skin, in situ malignancy, or curatively treated low-risk prostate cancer
* Known hypersensitivity to rituximab, bortezomib, boron, or any of the other agents used in this study
* Less than 14 days since prior investigational drugs
* Less than 4 weeks since prior bortezomib therapy (12 weeks for rituximab) and recovered from toxic effects prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-03; Primary Completion 2013-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne H. Blaes, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota Medical Center - Fairview, Minneapolis, Minnesota
  - Washington University School of Medicine - Oncology Division, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated Study Participants: Study participants receiving bortezomib and rituximab for post-transplant lymphoproliferative disorders (PTLD).
  Induction Therapy:
  rituximab: 375 mg/m^2 intravenously on Days 1,8, 15 and 22 bortezomib: 1.3 mg/m^2 intravenous bolus days 1, 8, 15 and 22 If complete response, start Maintenance Therapy. If partial response or stable disease, start Single Agent Bortezomib. If progressive disease, discontinue study treatment.
  Single Agent Bortezomib bortezomib: 1.3 mg/m^2 intravenous bolus days 1, 4, 8, 11 every 21 days for 4 cycles.
  If complete response or partial response, start Maintenance Therapy. If stable disease or progressive disease, discontinue study treatment.
  Maintenance Therapy:
  rituximab: 375 mg/m^2 intravenously on Days 1,8, 15 and 22 bortezomib: 1.3 mg/m^2 intravenous bolus days 1, 8, 15 and 22 Repeat every 6 months for a total of 4 cycles.
Period: Induction Therapy
Arm/Group | Treated Study Participants
Started | 3
Completed | 3
Not Completed | 0
Period: Maintenance Therapy
Arm/Group | Treated Study Participants
Started | 2 (One participant removed from study after completing induction therapy due to progressive disease.)
Completed | 1
Not Completed | 1
Not completed — concurrent illness | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treated Study Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Overall (Complete and Partial) Response Rates
Time Frame: Day 1 to 2 Years Post Treatment
Measure: Number; unit: participants
Arm/Group | Treated Study Participants
Number analyzed (Participants) | 3
participants | 2

2. Secondary Outcome: Remission Duration Among Patients Who Respond to Treatment
Time Frame: Day 1 to 8 Months Post Treatment
Population: Both of the participants who responded to treatment were in remission at last contact or death.
Measure: Median (Full Range); unit: months
Arm/Group | Treated Study Participants
Number analyzed (Participants) | 2
months | 45 [22 to 68]

3. Secondary Outcome: Time to Treatment Failure
Time Frame: Day 1 to Time of Disease Progression
Population: Two participants had a complete response at the time they completed the study and were not included in this outcome measure.
Measure: Number; unit: months
Arm/Group | Treated Study Participants
Number analyzed (Participants) | 1
months | 1

4. Secondary Outcome: Relapse-free Survival
Time Frame: at 2 years
Measure: Number; unit: participants
Arm/Group | Treated Study Participants
Number analyzed (Participants) | 3
participants | 2

5. Secondary Outcome: Overall Survival
Time Frame: at 2 years
Measure: Number; unit: participants
Arm/Group | Treated Study Participants
Number analyzed (Participants) | 3
participants | 1

ADVERSE EVENTS:
Arm/Group | Treated Study Participants
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treated Study Participants (N=3)
Fever (General disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Renal failure (Renal and urinary disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Myoclonus (Musculoskeletal and connective tissue disorders) | 1
Confusion (Nervous system disorders) | 1
Neuropathic pain (Nervous system disorders) | 1
Psychosis (Nervous system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Delerium (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treated Study Participants (N=3)
Aspartate aminotransferase increased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Fever (General disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Myoclonus (Musculoskeletal and connective tissue disorders) | 1
Confusion (Nervous system disorders) | 1
Neuropathic pain (Nervous system disorders) | 1
Psychosis (Nervous system disorders) | 1
Rectal bleeding (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue/malaise (General disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No